CLINICAL TRIAL: NCT02002923
Title: Pulmonary Vein Isolation Versus Botulinum Toxin Injection Plus Pulmonary Vein Isolation in Patients With Atrial Fibrillation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BT_AF+PVI
Record Dates: First submitted 2013-12-02; First posted 2013-12-06 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Paroxysmal Atrial Fibrillation; Persistent Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Botulinum Toxins

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PVI only (Active Comparator)
  Interventions: Procedure: Pulmonary vein isolation
- PVI+BT injection (Active Comparator)
  Interventions: Procedure: Pulmonary vein isolation; Drug: Botulinum Toxin

INTERVENTIONS:
Procedure: Pulmonary vein isolation — The left atrium (LA) and pulmonary veins (PVs) are explored through a transeptal approach. Real-time 3D LA maps are reconstructed by using a nonfluoroscopic navigation system. The ipsilateral left and right PVs are encircled in one lesion line by circumferential PV isolation. Radiofrequency energy is delivered at 43°C, 35 W, 0.5 cm away from the PV ostia at the anterior wall, and is reduced to 43°C, 30 W, 1 cm away from the PV ostia at the posterior wall, with a saline irrigation speed of 17 mL/min. Each lesion is ablated continuously until the local potential amplitude decreased by >80% or RF energy deliveries exceeded 40 s. The endpoint of circumferential PV isolation is PV isolation. Additional ablation lines are created by connecting the left inferior PV to the mitral annulus (mitral isthmus) and the roof of the LA between the two superior PVs. After the end of the procedure the implantable loop recorder is implanted in the parasternal area of the chest.
Drug: Botulinum Toxin — Transseptal puncture is performed by used standard endovascular approach. Injection of the botulinum toxin is performed in main anatomical zones of ganglionated plexuses of left atrium using Myostar catheter (Biosense Webster).
  Arms: PVI+BT injection

SUMMARY:
The investigators have conducted a prospective, double-blind, randomized study to assess the comparative safety and efficacy of two different treatment strategies, PVI only versus PVI plus BT injection, in patients with persistent and paroxysmal AF. Results were assessed after follow-up of at least 1 years with the use of an implanted monitoring device (IMD).

ELIGIBILITY:
Inclusion Criteria:

* Persistent and paroxysmal AF

Exclusion Criteria:

* congestive heart failure
* LV ejection fraction < 35%
* left atrial diameter > 60 mm

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Freedom of AF or other atrial arrhythmias | 1 year

SECONDARY OUTCOMES:
serious adverse events | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- State Research Institute of Circulation Pathology, Novosibirsk, Russia

REFERENCES:
- See also: State Research Institute of Circulation Pathology Official Site — http://meshalkin.ru